CLINICAL TRIAL: NCT03275311
Title: Epidemiological Strategy and Medical Economic (ESME) Research Program / Academic Real World Database: Evolution of the Therapeutic Care in Metastatic Breast Cancer Across the French Comprehensive Cancer Centers From 2008
Brief Title: Evolution of the Therapeutic Care in Metastatic Breast Cancer From 2008
Acronym: ESME-MBC
Status: Recruiting | Type: Observational
Sponsor: UNICANCER (Other)
Collaborators: Roche Pharma AG (Industry); Pierre Fabre Laboratories (Industry); Pfizer (Industry); AstraZeneca (Industry); Merck Sharp & Dohme LLC (Industry); Eisai Inc. (Industry); Daiichi Sankyo (Industry); Eli Lilly and Company (Industry); Gilead Sciences (Industry); Seagen Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: ESMEMBC
Record Dates: First submitted 2017-06-27; First posted 2017-09-07 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2024-04

CONDITIONS: Metastatic Breast Cancer
Keywords: metastatic breast cancer; observational study; survival; real world data; real life setting
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Epidemiological Strategy and Medical Economic (ESME) Breast cancer Database is a multicenter real life database using a retrospective data collection process across 18 French comprehensive cancer centers (FCCC) spread over 20 sites. This database compiles data from patient's electronic medical records (EMR).

DETAILED DESCRIPTION:
This database compiles existing data retrieved fromp patient's electronic medical records (EMR) across the 18 French comprehensive cancer centers spread over 20 sites. .

The database includes data related to patient demographics, tumor characteristics (diagnosis, histology, relapses, metastatic disease, etc.), treatments (dates, INN, route of administration, treatment protocols, reason for termination, etc.), and clinical events. Data is collected at each participating site by technicians who are specifically trained for the project using an electronic data collection (eDC) tool.

Data imported into the final database are controlled, recoded, and harmonized before import according to the data management plan. All coding procedures are predefined by the data manager. There is no transmission of individual data; all data are centralized within each center using a shared anonymous format. All data is exclusively obtained retrospectively; no attempts are made to recover non available data from the patient's medical record by contacting healthcare providers or patients.

Cases selected to enter the ESME MBC data platform fulfill specific criteria: (1) Male or female ≥18 years old (2) metastatic breast cancer (3) with first metastasis treated (either completely or partially) at a participating site from January 2008 onwards.Treatment strategies considered include radiotherapy, chemotherapy, targeted therapy and endocrine therapy.

ELIGIBILITY:
Inclusion criteria :

* 18 years old patient
* Patient receiving chemotherapy, targeted therapy, immunotherapy, radiation therapy and hormonotherapy in a French Comprehensive Cancer Center.

Exclusion criteria : None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients treated for a metastatic breast cancer in a French Comprehensive Cancer Center over the selection period.
Sampling Method: Non-Probability Sample
Enrollment: 40000 (Estimated)
Dates: Start 2014-07 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Describe the evolution of therapeutic care | baseline
  Patient characteristics, tumor characteristics and treatment patterns

SECONDARY OUTCOMES:
Describe the impact of therapeutic strategies on survival criteria | From date of diagnosis or first treatment until the date of date of death from any cause. Follow up until 2023.
  Overall survival
Describe the impact of therapeutic strategies on survival criteria | From date of diagnosis or first treatment until the date of first documented progression or date of death from any cause. Follow up until 2023.
  Progression free survival

CONTACTS AND LOCATIONS:
Overall Officials: Lise Bosquet, MsC, Study Director — UNICANCER
Locations (20):
- France (20):
  - Institut de Cancérologie de l'Ouest - Paul Papin, Angers
  - Institut Bergonié, Bordeaux
  - Centre François Baclesse, Caen
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges-François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - Centre Léon Bérard, Lyon
  - Institut Paoli-Calmettes, Marseille
  - Institut régional du Cancer Montpellier / Val d'Aurelle, Montpellier
  - Institut de Cancérologie de Lorraine, Nancy
  - Institut de cancérologie de l'Ouest - René Gauducheau, Nantes
  - Centre Antoine Lacassagne, Nice
  - Institut Curie, Paris
  - Institut Jean Godinot, Reims
  - Centre Eugène Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut Curie - Hôpital René Huguenin, Saint-Cloud
  - Centre Paul Strauss, Strasbourg
  - Institut Claudius Regaud, Toulouse
  - Institut Gustave Roussy, Villejuif

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Delaloge S, Perol D, Courtinard C, Brain E, Asselain B, Bachelot T, Debled M, Dieras V, Campone M, Levy C, Jacot W, Lorgis V, Veyret C, Dalenc F, Ferrero JM, Uwer L, Kerbrat P, Goncalves A, Mouret-Reynier MA, Petit T, Jouannaud C, Vanlemmens L, Chenuc G, Guesmia T, Robain M, Cailliot C. Paclitaxel plus bevacizumab or paclitaxel as first-line treatment for HER2-negative metastatic breast cancer in a multicenter national observational study. Ann Oncol. 2016 Sep;27(9):1725-32. doi: 10.1093/annonc/mdw260. Epub 2016 Jul 19. PMID 27436849
- [Result] Jacquet E, Lardy-Cleaud A, Pistilli B, Franck S, Cottu P, Delaloge S, Debled M, Vanlemmens L, Leheurteur M, Guizard AV, Laborde L, Uwer L, Jacot W, Berchery D, Desmoulins I, Ferrero JM, Perrocheau G, Courtinard C, Brain E, Chabaud S, Robain M, Bachelot T. Endocrine therapy or chemotherapy as first-line therapy in hormone receptor-positive HER2-negative metastatic breast cancer patients. Eur J Cancer. 2018 May;95:93-101. doi: 10.1016/j.ejca.2018.03.013. Epub 2018 Apr 11. PMID 29655061
- [Result] Gobbini E, Ezzalfani M, Dieras V, Bachelot T, Brain E, Debled M, Jacot W, Mouret-Reynier MA, Goncalves A, Dalenc F, Patsouris A, Ferrero JM, Levy C, Lorgis V, Vanlemmens L, Lefeuvre-Plesse C, Mathoulin-Pelissier S, Petit T, Uwer L, Jouannaud C, Leheurteur M, Lacroix-Triki M, Cleaud AL, Robain M, Courtinard C, Cailliot C, Perol D, Delaloge S. Time trends of overall survival among metastatic breast cancer patients in the real-life ESME cohort. Eur J Cancer. 2018 Jun;96:17-24. doi: 10.1016/j.ejca.2018.03.015. Epub 2018 Apr 13. PMID 29660596
- [Result] Cabel L, Carton M, Cheaib B, Pierga JY, Dalenc F, Mailliez A, Levy C, Jacot W, Debled M, Leheurteur M, Desmoulins I, Lefeuvre C, Goncalves A, Uwer L, Ferrero JM, Eymard JC, Petit T, Mouret-Reynier MA, Perrocheau G, Piot I, Perol D, Simon G, Lerebours F. Oral etoposide in heavily pre-treated metastatic breast cancer: results from the ESME cohort and comparison with other chemotherapy regimens. Breast Cancer Res Treat. 2019 Jan;173(2):397-406. doi: 10.1007/s10549-018-5017-2. Epub 2018 Oct 24. PMID 30357526
- [Result] Pons-Tostivint E, Kirova Y, Lusque A, Campone M, Geffrelot J, Mazouni C, Mailliez A, Pasquier D, Madranges N, Firmin N, Crouzet A, Goncalves A, Jankowski C, De La Motte Rouge T, Pouget N, de La Lande B, Mouttet-Boizat D, Ferrero JM, Uwer L, Eymard JC, Mouret-Reynier MA, Petit T, Robain M, Filleron T, Cailliot C, Dalenc F. Survival Impact of Locoregional Treatment of the Primary Tumor in De Novo Metastatic Breast Cancers in a Large Multicentric Cohort Study: A Propensity Score-Matched Analysis. Ann Surg Oncol. 2019 Feb;26(2):356-365. doi: 10.1245/s10434-018-6831-9. Epub 2018 Dec 11. PMID 30539492
- [Result] Delaloge S, Perol D, Robain M, Cailliot C. Reply to 'The potential and perils of observational studies' by M. Buyse et al. Ann Oncol. 2017 Feb 1;28(2):436-437. doi: 10.1093/annonc/mdw572. No abstract available. PMID 27831508
- [Result] Perol D, Robain M, Delaloge S, Cailliot C. Routinely collected data may usefully supplement randomised controlled data on treatment effects for mortality. BMJ. 2016 Dec 16;355:i6745. doi: 10.1136/bmj.i6745. No abstract available. PMID 27986716
- [Result] Petitjean A, Smith-Palmer J, Valentine W, Tehard B, Roze S. Cost-effectiveness of bevacizumab plus paclitaxel versus paclitaxel for the first-line treatment of HER2-negative metastatic breast cancer in specialist oncology centers in France. BMC Cancer. 2019 Feb 11;19(1):140. doi: 10.1186/s12885-019-5335-8. PMID 30744578
- [Result] Perol D, Robain M, Arveux P, Mathoulin-Pelissier S, Chamorey E, Asselain B, Berchery D, Gourgou S, Breton M, Delaine-Clisant S, Mons M, Dieras V, Carton M, Guizard AV, Laborde L, Laurent C, Loeb A, Mouret-Reynier MA, Parent D, Perrocheau G, Campion L, Velten M, Cailliot C, Ezzalfani M, Simon G. The ongoing French metastatic breast cancer (MBC) cohort: the example-based methodology of the Epidemiological Strategy and Medical Economics (ESME). BMJ Open. 2019 Feb 21;9(2):e023568. doi: 10.1136/bmjopen-2018-023568. PMID 30796119
- [Result] Jacot W, Heudel PE, Fraisse J, Gourgou S, Guiu S, Dalenc F, Pistilli B, Campone M, Levy C, Debled M, Leheurteur M, Chaix M, Lefeuvre C, Goncalves A, Uwer L, Ferrero JM, Eymard JC, Petit T, Mouret-Reynier MA, Courtinard C, Cottu P, Robain M, Mailliez A. Real-life activity of eribulin mesylate among metastatic breast cancer patients in the multicenter national observational ESME program. Int J Cancer. 2019 Dec 15;145(12):3359-3369. doi: 10.1002/ijc.32402. Epub 2019 Jun 20. PMID 31087564
- [Result] Le Saux O, Lardy-Cleaud A, Frank S, Debled M, Cottu PH, Pistilli B, Vanlemmens L, Leheurteur M, Levy C, Laborde L, Uwer L, D'hondt V, Berchery D, Lorgis V, Ferrero JM, Perrocheau G, Courtinard C, Mouret-Reynier MA, Velten M, Breton M, Parent D, Chabaud S, Robain M, Bachelot T. Assessment of the efficacy of successive endocrine therapies in hormone receptor-positive and HER2-negative metastatic breast cancer: a real-life multicentre national study. Eur J Cancer. 2019 Sep;118:131-141. doi: 10.1016/j.ejca.2019.06.014. Epub 2019 Jul 19. PMID 31330488
- [Result] Gougis P, Carton M, Tchokothe C, Campone M, Dalenc F, Mailliez A, Levy C, Jacot W, Debled M, Leheurteur M, Bachelot T, Hennequin A, Perrin C, Goncalves A, Uwer L, Eymard JC, Petit T, Mouret-Reynier MA, Chamorey E, Simon G, Saghatchian M, Cailliot C, Le Tourneau C. CineBreast-factors influencing the time to first metastatic recurrence in breast cancer: Analysis of real-life data from the French ESME MBC database. Breast. 2020 Feb;49:17-24. doi: 10.1016/j.breast.2019.10.004. Epub 2019 Oct 19. PMID 31675683
- [Result] Darlix A, Louvel G, Fraisse J, Jacot W, Brain E, Debled M, Mouret-Reynier MA, Goncalves A, Dalenc F, Delaloge S, Campone M, Augereau P, Ferrero JM, Levy C, Fumet JD, Lecouillard I, Cottu P, Petit T, Uwer L, Jouannaud C, Leheurteur M, Dieras V, Robain M, Chevrot M, Pasquier D, Bachelot T. Impact of breast cancer molecular subtypes on the incidence, kinetics and prognosis of central nervous system metastases in a large multicentre real-life cohort. Br J Cancer. 2019 Dec;121(12):991-1000. doi: 10.1038/s41416-019-0619-y. Epub 2019 Nov 13. PMID 31719684
- [Result] Pasquier D, Darlix A, Louvel G, Fraisse J, Jacot W, Brain E, Petit A, Mouret-Reynier MA, Goncalves A, Dalenc F, Deluche E, Fresnel JS, Augereau P, Ferrero JM, Geffrelot J, Fumet JD, Lecouillard I, Cottu P, Petit T, Uwer L, Jouannaud C, Leheurteur M, Dieras V, Robain M, Mouttet-Audouard R, Bachelot T, Courtinard C. Treatment and outcomes in patients with central nervous system metastases from breast cancer in the real-life ESME MBC cohort. Eur J Cancer. 2020 Jan;125:22-30. doi: 10.1016/j.ejca.2019.11.001. Epub 2019 Dec 10. PMID 31835235
- [Result] Deluche E, Antoine A, Bachelot T, Lardy-Cleaud A, Dieras V, Brain E, Debled M, Jacot W, Mouret-Reynier MA, Goncalves A, Dalenc F, Patsouris A, Ferrero JM, Levy C, Lorgis V, Vanlemmens L, Lefeuvre-Plesse C, Mathoulin-Pelissier S, Petit T, Uwer L, Jouannaud C, Leheurteur M, Lacroix-Triki M, Courtinard C, Perol D, Robain M, Delaloge S. Contemporary outcomes of metastatic breast cancer among 22,000 women from the multicentre ESME cohort 2008-2016. Eur J Cancer. 2020 Apr;129:60-70. doi: 10.1016/j.ejca.2020.01.016. Epub 2020 Mar 2. PMID 32135312
- [Result] Pons-Tostivint E, Kirova Y, Lusque A, Campone M, Geffrelot J, Rivera S, Mailliez A, Pasquier D, Madranges N, Firmin N, Crouzet A, Goncalves A, Jankowski C, De La Motte Rouge T, Pouget N, De La Lande B, Mouttet-Boizat D, Ferrero JM, Uwer L, Eymard JC, Mouret-Reynier MA, Petit T, Courtinard C, Filleron T, Robain M, Dalenc F. Radiation therapy to the primary tumor for de novo metastatic breast cancer and overall survival in a retrospective multicenter cohort analysis. Radiother Oncol. 2020 Apr;145:109-116. doi: 10.1016/j.radonc.2019.12.019. Epub 2020 Jan 10. PMID 31931289
- [Result] Heudel P, Delaloge S, Parent D, Madranges N, Levy C, Dalenc F, Brain E, Uwer L, D'Hondt V, Augereau P, Mailliez A, Perrin C, Frenel JS, Sablin MP, Mouret-Reynier MA, Vermeulin T, Eymard JC, Petit T, Ferrero JM, Ilie S, Goncalves A, Chenuc G, Robain M, Simon G, Perol D. Real-world Evaluation of Oral Vinorelbine in the Treatment of Metastatic Breast Cancer: An ESME-MBC Study. Anticancer Res. 2020 Jul;40(7):3905-3913. doi: 10.21873/anticanres.14381. PMID 32620631
- [Result] Frasca M, Sabathe C, Delaloge S, Galvin A, Patsouris A, Levy C, Mouret-Reynier MA, Desmoulins I, Vanlemmens L, Bachelot T, Goncalves A, Perotin V, Uwer L, Frenel JS, Ferrero JM, Bouleuc C, Eymard JC, Dieras V, Leheurteur M, Petit T, Dalenc F, Jaffre A, Chevrot M, Courtinard C, Mathoulin-Pelissier S. Palliative care delivery according to age in 12,000 women with metastatic breast cancer: Analysis in the multicentre ESME-MBC cohort 2008-2016. Eur J Cancer. 2020 Sep;137:240-249. doi: 10.1016/j.ejca.2020.07.007. Epub 2020 Aug 14. PMID 32805641
- [Result] Frank S, Carton M, Dubot C, Campone M, Pistilli B, Dalenc F, Mailliez A, Levy C, D'Hondt V, Debled M, Vermeulin T, Coudert B, Perrin C, Goncalves A, Uwer L, Ferrero JM, Eymard JC, Petit T, Mouret-Reynier MA, Patsouris A, Guesmia T, Bachelot T, Robain M, Cottu P. Impact of age at diagnosis of metastatic breast cancer on overall survival in the real-life ESME metastatic breast cancer cohort. Breast. 2020 Aug;52:50-57. doi: 10.1016/j.breast.2020.04.009. Epub 2020 Apr 23. PMID 32380440
- [Result] Saleh K, Carton M, Dieras V, Heudel PE, Brain E, D'Hondt V, Mailliez A, Patsouris A, Mouret-Reynier MA, Goncalves A, Ferrero JM, Petit T, Emile G, Uwer L, Debled M, Dalenc F, Jouannaud C, Ladoire S, Leheurteur M, Cottu P, Veron L, Savignoni A, Courtinard C, Robain M, Delaloge S, Deluche E. Impact of body mass index on overall survival in patients with metastatic breast cancer. Breast. 2021 Feb;55:16-24. doi: 10.1016/j.breast.2020.11.014. Epub 2020 Dec 1. PMID 33307392
- [Result] Sirieix J, Fraisse J, Mathoulin-Pelissier S, Leheurteur M, Vanlemmens L, Jouannaud C, Dieras V, Levy C, Ung M, Mouret-Reynier MA, Petit T, Coudert B, Brain E, Pistilli B, Ferrero JM, Goncalves A, Uwer L, Patsouris A, Tredan O, Courtinard C, Gourgou S, Frenel JS. Management and outcome of male metastatic breast cancer in the national multicenter observational research program Epidemiological Strategy and Medical Economics (ESME). Ther Adv Med Oncol. 2020 Dec 23;12:1758835920980548. doi: 10.1177/1758835920980548. eCollection 2020. PMID 33488779
- [Result] Bertho M, Fraisse J, Patsouris A, Cottu P, Arnedos M, Perol D, Jaffre A, Goncalves A, Lebitasy MP, D'Hondt V, Dalenc F, Ferrero JM, Levy C, Dabakuyo S, Rouzier R, Penault-Llorca F, Uwer L, Eymard JC, Breton M, Chevrot M, Thureau S, Petit T, Simon G, Frenel JS. Real-life prognosis of 5041 bone-only metastatic breast cancer patients in the multicenter national observational ESME program. Ther Adv Med Oncol. 2021 Jan 21;13:1758835920987657. doi: 10.1177/1758835920987657. eCollection 2021. PMID 33613700
- [Result] Cabel L, Carton M, Pistilli B, Dalenc F, Vanlemnens L, Levy C, Jacot W, Debled M, Loeb A, Hennequin A, De la Motte Rouge T, Laborde L, Laurent C, Chamorey E, Parent D, Petit T, Mouret-Reynier MA, Campone M, Perrocheau G, Labreveux C, Bachelot T, Robain M, Lerebours F. Outcome beyond third-line chemotherapy for metastatic triple-negative breast cancer in the French ESME program. Breast. 2021 Apr;56:18-25. doi: 10.1016/j.breast.2021.01.006. Epub 2021 Jan 30. PMID 33561617
- [Result] Hotton J, Lusque A, Leufflen L, Campone M, Levy C, Honart JF, Mailliez A, Debled M, Gutowski M, Leheurteur M, Goncalves A, Jankowski C, Guillermet S, Bachelot T, Ferrero JM, Eymard JC, Petit T, Pouget N, de La Lande B, Frenel JS, Villacroux O, Simon G, Pons-Tostivint E, Marchai F. Early Locoregional Breast Surgery and Survival in de novo Metastatic Breast Cancer in the Multicenter National ESME Cohort. Ann Surg. 2023 Jan 1;277(1):e153-e161. doi: 10.1097/SLA.0000000000004767. Epub 2021 Feb 1. PMID 33534229
- [Result] Annonay M, Gauquelin L, Geiss R, Ung M, Cristol-Dalstein L, Mouret-Reynier MA, Goncalves A, Abadie-Lacourtoisie S, Francois E, Perrin C, Le Fel J, Lorgis V, Servent V, Uwer L, Jouannaud C, Leheurteur M, Joly F, Campion L, Courtinard C, Villacroux O, Petit T, Soubeyran P, Terret C, Bellera C, Brain E, Delaloge S. Treatment and outcomes of older versus younger women with HER2-positive metastatic breast cancer in the real-world national ESME database. Breast. 2021 Dec;60:138-146. doi: 10.1016/j.breast.2021.09.011. Epub 2021 Oct 1. PMID 34624756
- [Result] Carausu M, Carton M, Darlix A, Pasquier D, Leheurteur M, Debled M, Mouret-Reynier MA, Goncalves A, Dalenc F, Verret B, Campone M, Augereau P, Ferrero JM, Levy C, Fumet JD, Lefeuvre-Plesse C, Petit T, Uwer L, Jouannaud C, Larrouquere L, Chevrot M, Courtinard C, Cabel L. Breast cancer patients treated with intrathecal therapy for leptomeningeal metastases in a large real-life database. ESMO Open. 2021 Jun;6(3):100150. doi: 10.1016/j.esmoop.2021.100150. Epub 2021 May 10. PMID 33984675
- [Result] Corbaux P, Lardy-Cleaud A, Alexandre M, Fontanilles M, Levy C, Viansone AA, Mailliez A, Debled M, Goncalves A, Le Du F, Lerebours F, Ferrero JM, Eymard JC, Mouret-Reynier MA, Petit T, Frenel JS, Dalenc F, Courtinard C, Chaix M, Bachelot T. Progression-free survival on endocrine therapy, before or after chemotherapy, in hormone receptor-positive HER2-negative metastatic breast cancer. Breast Cancer Res Treat. 2022 Jan;191(1):191-207. doi: 10.1007/s10549-021-06382-6. Epub 2021 Oct 23. PMID 34687411
- [Result] Dano D, Lardy-Cleaud A, Monneur A, Quenel-Tueux N, Levy C, Mouret-Reynier MA, Coudert B, Mailliez A, Ferrero JM, Guiu S, Campone M, de La Motte Rouge T, Petit T, Pistilli B, Dalenc F, Simon G, Lerebours F, Chabaud S, Bertucci F, Goncalves A. Metastatic inflammatory breast cancer: survival outcomes and prognostic factors in the national, multicentric, and real-life French cohort (ESME). ESMO Open. 2021 Aug;6(4):100220. doi: 10.1016/j.esmoop.2021.100220. Epub 2021 Jul 22. PMID 34303929
- [Result] Ezzalfani M, Porcher R, Savignoni A, Delaloge S, Filleron T, Robain M, Perol D; ESME Group. Addressing the issue of bias in observational studies: Using instrumental variables and a quasi-randomization trial in an ESME research project. PLoS One. 2021 Sep 15;16(9):e0255017. doi: 10.1371/journal.pone.0255017. eCollection 2021. PMID 34525119
- [Result] Gaillard T, Carton M, Mailliez A, Desmoulins I, Mouret-Reynier MA, Petit T, Leheurteur M, Dieras V, Ferrero JM, Uwer L, Guiu S, Goncalves A, Levy C, Debled M, Dalenc F, Patsouris A, Bachelot T, Eymard JC, Chevrot M, Conversano A, Robain M, Hequet D. De novo metastatic breast cancer in patients with a small locoregional tumour (T1-T2/N0): Characteristics and prognosis. Eur J Cancer. 2021 Nov;158:181-188. doi: 10.1016/j.ejca.2021.09.021. Epub 2021 Oct 21. PMID 34689042
- [Result] Grinda T, Antoine A, Jacot W, Blaye C, Cottu PH, Dieras V, Dalenc F, Goncalves A, Debled M, Patsouris A, Mouret-Reynier MA, Mailliez A, Clatot F, Levy C, Ferrero JM, Desmoulins I, Uwer L, Petit T, Jouannaud C, Lacroix-Triki M, Deluche E, Robain M, Courtinard C, Bachelot T, Brain E, Perol D, Delaloge S. Evolution of overall survival and receipt of new therapies by subtype among 20 446 metastatic breast cancer patients in the 2008-2017 ESME cohort. ESMO Open. 2021 Jun;6(3):100114. doi: 10.1016/j.esmoop.2021.100114. Epub 2021 Apr 23. PMID 33895695
- [Result] Grinda T, Joyon N, Lusque A, Lefevre S, Arnould L, Penault-Llorca F, Macgrogan G, Treilleux I, Vincent-Salomon A, Haudebourg J, Maran-Gonzalez A, Charafe-Jauffret E, Courtinard C, Franchet C, Verriele V, Brain E, Tas P, Blanc-Fournier C, Leroux A, Loussouarn D, Berghian A, Brabencova E, Ghnassia JP, Scoazec JY, Delaloge S, Filleron T, Lacroix-Triki M. Phenotypic discordance between primary and metastatic breast cancer in the large-scale real-life multicenter French ESME cohort. NPJ Breast Cancer. 2021 Apr 16;7(1):41. doi: 10.1038/s41523-021-00252-6. PMID 33863896
- [Result] Bringuier M, Carton M, Levy C, Patsouris A, Pasquier D, Debled M, Rigal O, Jacot W, Goncalves A, Desmoulins I, De La Motte Rouge T, Bachelot T, Ferrero JM, Eymard JC, Ung M, Mouret-Reynier MA, Petit T, Chevrot M, Uwer L, Courtinard C, Frenel JS, Vianzone A, Baldini C. Enrollment of older metastatic breast cancer patients in first-line clinical trials: 9-year experience of the large-scale real-life multicenter French ESME cohort. Breast Cancer Res Treat. 2022 Feb;191(3):577-587. doi: 10.1007/s10549-021-06467-2. Epub 2022 Jan 5. PMID 34984582
- [Result] Carausu M, Carton M, Cabel L, Patsouris A, Levy C, Verret B, Pasquier D, Debled M, Goncalves A, Desmoulins I, Lecouillard I, Bachelot T, Ferrero JM, Eymard JC, Mouret-Reynier MA, Chevrot M, De Maio E, Uwer L, Frenel JS, Leheurteur M, Petit T, Darlix A, Bozec L. Clinicopathological characteristics and prognosis of breast cancer patients with isolated central nervous system metastases in the multicentre ESME database. Ther Adv Med Oncol. 2022 Feb 26;14:17588359221077082. doi: 10.1177/17588359221077082. eCollection 2022. PMID 35237352
- [Result] Dalenc F, Lusque A, De La Motte Rouge T, Pistilli B, Brain E, Pasquier D, Debled M, Thery JC, Goncalves A, Desmoulins I, Levy C, Uwer L, Ferrero JM, Eymard JC, Mouret-Reynier MA, Patsouris A, Frenel JS, Petit T, Chevrot M, Bachelot T, Guiu S. Impact of lobular versus ductal histology on overall survival in metastatic breast cancer: a French retrospective multicentre cohort study. Eur J Cancer. 2022 Mar;164:70-79. doi: 10.1016/j.ejca.2021.12.031. Epub 2022 Feb 14. PMID 35176614
- [Result] Mallet A, Lusque A, Levy C, Pistilli B, Brain E, Pasquier D, Debled M, Thery JC, Goncalves A, Desmoulins I, De La Motte Rouge T, Faure C, Ferrero JM, Eymard JC, Mouret-Reynier MA, Patsouris A, Cottu P, Dalenc F, Petit T, Payen O, Uwer L, Guiu S, Frenel JS. Real-world evidence of the management and prognosis of young women (⩽40 years) with de novo metastatic breast cancer. Ther Adv Med Oncol. 2022 Jan 21;14:17588359211070362. doi: 10.1177/17588359211070362. eCollection 2022. PMID 35082924
- [Result] Moinard-Butot F, Saint-Martin C, Pflumio C, Carton M, Jacot W, Cottu PH, Dieras V, Dalenc F, Goncalves A, Debled M, Patsouris A, Mouret-Reynier MA, Vanlemmens L, Leheurteur M, Emile G, Ferrero JM, Desmoulins I, Uwer L, Eymard JC, Cheaib B, Courtinard C, Bachelot T, Chevrot M, Petit T. Efficacy of trastuzumab emtansine (T-DM1) and lapatinib after dual HER2 inhibition with trastuzumab and pertuzumab in patient with metastatic breast cancer: Retrospective data from a French multicenter real-life cohort. Breast. 2022 Jun;63:54-60. doi: 10.1016/j.breast.2022.03.004. Epub 2022 Mar 11. PMID 35299035
- [Result] Vasseur A, Carton M, Guiu S, Augereau P, Uwer L, Mouret-Reynier MA, Levy C, Eymard JC, Ferrero JM, Leheurteur M, Goncalves A, Robert M, De La Motte Rouge T, Bachelot T, Petit T, Debled M, Grinda T, Desmoulins I, Vanlemmens L, Nicolai V, Simon G, Cabel L. Efficacy of taxanes rechallenge in first-line treatment of early metastatic relapse of patients with HER2-negative breast cancer previously treated with a (neo)adjuvant taxanes regimen: A multicentre retrospective observational study. Breast. 2022 Oct;65:136-144. doi: 10.1016/j.breast.2022.07.014. Epub 2022 Aug 4. PMID 35944353
- [Result] Jacot W, Lusque A, Vicier C, Mailliez A, de La Motte Rouge T, Cabel L, Levy C, Patsouris A, Desmoulins I, Uwer L, Thery JC, Robain M, Caron O, Tredan O, Filleron T, Frenel JS, Delaloge S. Outcomes of patients with HER2-negative metastatic breast cancer after platinum- and non-platinum-based first-line chemotherapy among patients with and without pathogenic germline BRCA1/2 mutations. Br J Cancer. 2022 Nov;127(11):1963-1973. doi: 10.1038/s41416-022-02003-1. Epub 2022 Oct 7. PMID 36207609
- [Result] Mailliez A, D'Hondt V, Lusque A, Caron O, Cabel L, Goncalves A, Debled M, Gladieff L, Ferrero JM, Petit T, Mouret-Reynier MA, Eymard JC, Levy C, Uwer L, Leheurteur M, Desmoulins I, Bachelot T, Frenel JS, de la Motte Rouge T, Simon G, Jacot W, Delaloge S. Survival outcomes of metastatic breast cancer patients by germline BRCA1/2 status in a large multicenter real-world database. Int J Cancer. 2023 Mar 1;152(5):921-931. doi: 10.1002/ijc.34304. Epub 2022 Oct 8. PMID 36161271
- [Result] de Calbiac O, Lusque A, Mailliez A, Bachelot T, Uwer L, Mouret-Reynier MA, Emile G, Jouannaud C, Goncalves A, Patsouris A, Dieras V, Leheurteur M, Petit T, Cottu P, Ferrero JM, D'Hondt V, Desmoulins I, Mourato-Ribeiro J, Martin AL, Frenel JS. Comparison of Management and Outcomes in ERBB2-Low vs ERBB2-Zero Metastatic Breast Cancer in France. JAMA Netw Open. 2022 Sep 1;5(9):e2231170. doi: 10.1001/jamanetworkopen.2022.31170. PMID 36107428
- [Result] Carausu M, Carton M, Dieras V, Petit T, Guiu S, Goncalves A, Augereau P, Ferrero JM, Levy C, Ung M, Desmoulins I, Debled M, Bachelot T, Pistilli B, Frenel JS, Mailliez A, Chevrot M, Cabel L. Association of Endocrine Therapy for HR+/ERBB2+ Metastatic Breast Cancer With Survival Outcomes. JAMA Netw Open. 2022 Dec 1;5(12):e2247154. doi: 10.1001/jamanetworkopen.2022.47154. PMID 36520434
- [Result] Collet L, Eberst L, Ludovic G, Debled M, Hrab L, Mouret-Reynier MA, Desmoulins I, Goncalves A, Campone M, Ferrero JM, Brain E, Uwer L, Eymard JC, Dieras V, Simon G, Leheurteur M, Dalenc F, Vanlemmens L, Darlix A, Arnedos M, Bachelot T. Clinical outcome of patients with isolated central nervous system progression on first-line pertuzumab and trastuzumab treatment for HER2-positive metastatic breast cancer in a real-life cohort. Breast Cancer. 2023 Mar;30(2):329-341. doi: 10.1007/s12282-022-01427-0. Epub 2023 Jan 11. PMID 36630013
- [Result] Francois-Martin H, Lardy-Cleaud A, Pistilli B, Levy C, Dieras V, Frenel JS, Guiu S, Mouret-Reynier MA, Mailliez A, Eymard JC, Petit T, Ung M, Desmoulins I, Augereau P, Bachelot T, Uwer L, Debled M, Ferrero JM, Clatot F, Goncalves A, Chevrot M, Chabaud S, Cottu P. Long-Term Results with Everolimus in Advanced Hormone Receptor Positive Breast Cancer in a Multicenter National Real-World Observational Study. Cancers (Basel). 2023 Feb 13;15(4):1191. doi: 10.3390/cancers15041191. PMID 36831532
- [Result] Courtinard C, Gourgou S, Jacot W, Carton M, Guerin O, Vacher L, Bertaut A, Le Deley MC, Perol D, Marino P, Levy C, Uwer L, Perrocheau G, Schiappa R, Bachelot F, Parent D, Breton M, Petit T, Filleron T, Loeb A, Mathoulin-Pelissier S, Robain M, Delaloge S, Bellera C. Association between progression-free survival and overall survival in women receiving first-line treatment for metastatic breast cancer: evidence from the ESME real-world database. BMC Med. 2023 Mar 8;21(1):87. doi: 10.1186/s12916-023-02754-5. PMID 36882736
- [Result] Frenel JS, Lusque A, Delaloge S, Ferrero JM, Bachelot T, Desmoulins I, Levy C, Eymard JC, Goncalves A, Patsouris A, Reynier MAM, Thery MJ, Petit T, Cabel L, Uwer L, Debled M, Chevrot M, Mailliez A, Jacot W, de La Motte Rouge T. Efficacy of front-line treatment for hormone receptor-positive HER2-negative metastatic breast cancer with germline BRCA1/2 mutation. Br J Cancer. 2023 Jun;128(11):2072-2080. doi: 10.1038/s41416-023-02248-4. Epub 2023 Apr 3. PMID 37012318
- [Result] Antoine A, Perol D, Robain M, Delaloge S, Lasset C, Drouet Y. Target trial emulation to assess real-world efficacy in the Epidemiological Strategy and Medical Economics metastatic breast cancer cohort. J Natl Cancer Inst. 2023 Aug 8;115(8):971-980. doi: 10.1093/jnci/djad092. PMID 37220893
- [Result] Grinda T, Antoine A, Jacot W, Cottu PH, de la Motte Rouge T, Frenel JS, Mailliez A, Dalenc F, Goncalves A, Clatot F, Mouret Reynier MA, Levy C, Ferrero JM, Desmoulins I, Uwer L, Petit T, Jouannaud C, Arnedos M, Chevrot M, Courtinard C, Tredan O, Brain E, Perol D, Pistilli B, Delaloge S. Real-world clinical and survival outcomes of patients with early relapsed triple-negative breast cancer from the ESME national cohort. Eur J Cancer. 2023 Aug;189:112935. doi: 10.1016/j.ejca.2023.05.023. Epub 2023 Jun 7. PMID 37385070
- [Result] Le Du F, Carton M, Bachelot T, Saghatchian M, Pistilli B, Brain E, Loirat D, Vanlemmens L, Vermeulin T, Emile G, Goncalves A, Ung M, Robert M, Jaffre A, Desmoulins I, Jouannaud C, Uwer L, Marc Ferrero J, Mouret-Reynier MA, Jacot W, Chevrot M, Delaloge S, Dieras V. Real-World Impact of Adjuvant Anti-HER2 Treatment on Characteristics and Outcomes of Women With HER2-Positive Metastatic Breast Cancer in the ESME Program. Oncologist. 2023 Oct 3;28(10):e867-e876. doi: 10.1093/oncolo/oyad137. PMID 37589218
- [Result] Galvin A, Courtinard C, Bouteiller F, Gourgou S, Dalenc F, Jacot W, Arnedos M, Bailleux C, Dieras V, Petit T, Emile G, Dubray-Longeras P, Frenel JS, Bachelot T, Mailliez A, Brain E, Desmoulins I, Massard V, Patsouris A, Goncalves A, Grinda T, Delaloge S, Bellera C. First-line real-world treatment patterns and survival outcomes in women younger or older than 40 years with metastatic breast cancer in the real-life multicenter French ESME cohort. Eur J Cancer. 2024 Jan;196:113422. doi: 10.1016/j.ejca.2023.113422. Epub 2023 Nov 10. PMID 37977105
- [Result] Epaillard N, Lusque A, Jacot W, Mailliez A, Bachelot T, Arnedos M, Le Du F, Brain E, Ferrero JM, Massard V, Desmoulins I, Mouret-Reynier MA, Levy C, Goncalves A, Leheurteur M, Petit T, Filleron T, Bosquet L, Pistilli B, Frenel JS. Incidence and outcome of brain and/or leptomeningeal metastases in HER2-low metastatic breast cancer in the French ESME cohort. ESMO Open. 2024 May;9(5):103447. doi: 10.1016/j.esmoop.2024.103447. Epub 2024 May 3. PMID 38703431
- [Result] Courtinard C, Barbet V, Schiappa R, Pilleul F, Michiels S, Dabakuyo S, Gourgou S, Jaffre A, Asselain B, Bosquet L, Dunton K, Rosenlund M, Liang Z, Cathcart J, Delaloge S. Real-word effectiveness of post-trastuzumab emtansine treatment for human epidermal growth factor. Receptor 2-positive metastatic breast cancer: a multicenter, matched cohort analysis from the Epidermology Strategy and Medical Economics database (2008-2018). Real-World Data and Digital Oncology. 2024 https://doi.org/10.1016/j.esmorw.2024.100043
- [Result] Antoine A, Perol D, Robain M, Bachelot T, Choquet R, Jacot W, Ben Hadj Yahia B, Grinda T, Delaloge S, Lasset C, Drouet Y. Assessing the real-world effectiveness of 8 major metastatic breast cancer drugs using target trial emulation. Eur J Cancer. 2024 Dec;213:115072. doi: 10.1016/j.ejca.2024.115072. Epub 2024 Oct 22. PMID 39476445